CLINICAL TRIAL: NCT04495478
Title: A Single-Dose Study in Healthy Participants to Characterize Ramucirumab Pharmacokinetics and Investigate Injection Site Reactions Following an Intravenous Infusion or Subcutaneous Administration of Ramucirumab
Brief Title: A Study of Ramucirumab (LY3009806) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17748; I4T-MC-JVDT (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-07-30; First posted 2020-07-31 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo - Intravenous (IV) (Experimental): Participants received single dose of placebo administered IV.
  Interventions: Drug: Placebo - IV
- 350 mg Ramucirumab IV (Placebo Comparator): Participants received single 350 milligram (mg) ramucirumab administered as a 60-minute intravenous infusion at a concentration of 10 milligram per millilitre (mg/mL) as one 35 mL infusion.
  Interventions: Drug: Ramucirumab - IV
- Placebo - Subcutaneous (SC) (Experimental): Participants received single dose of placebo administered SC.
  Interventions: Drug: Placebo - SC
- 350 mg Ramucirumab SC (1x2 mL) (Placebo Comparator): Participants received single 350 mg ramucirumab SC administered at a concentration of 175 mg/mL as one 2 mL injection.
  Interventions: Drug: Ramucirumab - SC
- 350 mg Ramucirumab SC (2x2 mL) (Experimental): Participants received single 350 mg ramucirumab SC administered at a concentration of 87.5 mg/mL as two 2 mL injections.
  Interventions: Drug: Ramucirumab - SC
- 350 mg Ramucirumab SC (2x1 mL) (Experimental): Participants received single 350 mg ramucirumab SC administered at a concentration of 175 mg/mL as two 1 mL injections.
  Interventions: Drug: Ramucirumab - SC
- 700 mg Ramucirumab SC (2x2 mL) (Experimental): Participants received single 700 mg ramucirumab SC administered at a concentration of 175 mg/mL as two 2 mL injections.
  Interventions: Drug: Ramucirumab - SC

INTERVENTIONS:
Drug: Ramucirumab - IV — Administered IV.
  Other Names: LY3009806
  Arms: 350 mg Ramucirumab IV
Drug: Placebo - IV — Administered IV.
  Arms: Placebo - Intravenous (IV)
Drug: Ramucirumab - SC — Administered SC.
  Other Names: LY3009806
  Arms: 350 mg Ramucirumab SC (1x2 mL); 350 mg Ramucirumab SC (2x1 mL); 350 mg Ramucirumab SC (2x2 mL); 700 mg Ramucirumab SC (2x2 mL)
Drug: Placebo - SC — Administered SC.
  Arms: Placebo - Subcutaneous (SC)

SUMMARY:
This study evaluates a new formulation of ramucirumab, a drug approved for several types of cancer.

In this study of healthy participants, a small amount of ramucirumab will be given by injection either into a vein or just under the skin. Study doctors will measure the amount of ramucirumab in the bloodstream.

Side effects and tolerability will be documented. The study will last for about 16 weeks for each participant, including screening and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until study completion)
* Have a body weight greater than or equal to (≥)70 kilograms (kg) and body mass index (BMI) of 18 to 32 kilogram per square meter (kg/m ²), inclusive
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 500 milliliters (mL) within the previous 30 days of study screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo IV: Participants received single dose of placebo administered Intravenously (IV).
- Placebo SC: Participants received single dose of placebo administered subcutaneously (SC).
Period: Overall Study
Arm/Group | Placebo IV | 350 mg Ramucirumab IV | Placebo SC | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL)
Started | 3 | 7 | 12 | 7 | 7 | 7 | 7
Received at Least One Dose of Study Drug | 3 | 7 | 12 | 7 | 7 | 7 | 7
Completed | 3 | 6 | 12 | 6 | 6 | 7 | 7
Not Completed | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo IV: Participants received single dose of placebo administered IV.
- 350 mg Ramucirumab IV: Participants received single 350 mg ramucirumab administered as a 60-minute intravenous infusion at a concentration of 10 mg/mL as one 35 mL infusion.
- Placebo SC: Participants received single dose of placebo administered SC.
- Total: Total of all reporting groups
Arm/Group | Placebo IV | 350 mg Ramucirumab IV | Placebo SC | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL) | Total
Number analyzed (Participants) | 3 | 7 | 12 | 7 | 7 | 7 | 7 | 50
Age, Continuous [Median (Full Range); unit: years] | 34 [28 to 53] | 35 [20 to 54] | 37 [21 to 58] | 51 [24 to 59] | 46 [26 to 56] | 39 [21 to 60] | 41 [22 to 53] | 40 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 2 | 2 | 0 | 1 | 9
  Male | 3 | 5 | 10 | 5 | 5 | 7 | 6 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 7 | 4 | 4 | 2 | 1 | 23
  Not Hispanic or Latino | 1 | 4 | 5 | 3 | 3 | 5 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 0 | 2 | 2 | 2 | 12
  White | 2 | 4 | 8 | 6 | 5 | 5 | 5 | 35
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 7 | 12 | 7 | 7 | 7 | 7 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any adverse event from this study that results in 1 of the following: Death, initial or prolonged inpatient hospitalization, a life-threatening experience (that is, risk of death), persistent or significant disability/incapacity, congenital anomaly/birth defect, Important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent 1 of the other outcomes listed in the definition above. The number of participants with one or more SAEs considered by the investigator to be related to study drug administration is reported. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Time Frame: Baseline through Day 90
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | 350 mg Ramucirumab IV | Placebo SC | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL)
Number analyzed (Participants) | 3 | 7 | 12 | 7 | 7 | 7 | 7
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Injection Site Reactions (ISRs) Following Subcutaneous (SC) Administration of Study Drug
Description: Number of participants showing ISRs when the drug was administered subcutaneously were reported.
Time Frame: Day 1 Predose through Day 90
Population: All participants who received at least one dose of study drug subcutaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL)
Number analyzed (Participants) | 12 | 7 | 7 | 7 | 7
Participants | 3 | 3 | 2 | 1 | 1

3. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Ramucirumab
Description: PK: AUC[0-∞] of Ramucirumab.
Time Frame: 1, 8, 24, 48, 72, 96, 120, 144, 168, 264, 336, 504 hours post-dose
Population: All participants who received at least one dose of ramucirumab and had sufficient evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter (h*μg/mL)
Arm/Group | 350 mg Ramucirumab IV | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL)
Number analyzed (Participants) | 7 | 5 | 7 | 6 | 7
hour*microgram per milliliter (h*μg/mL) | 18700 (19) | 5250 (48) | 5140 (76) | 6350 (57) | 14200 (76)

4. Primary Outcome: PK: Maximum Concentration (Cmax) of Ramucirumab
Description: PK: Cmax of Ramucirumab
Time Frame: 1, 8, 24, 48, 72, 96, 120, 144, 168, 264, 336, 504 hours post-dose
Population: All participants who received at least one dose of ramucirumab and had sufficient evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 350 mg Ramucirumab IV | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL)
Number analyzed (Participants) | 7 | 6 | 7 | 7 | 7
μg/mL | 116 (11) | 24 (56) | 20.2 (63) | 21 (66) | 46.7 (44)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 90
Description: All participants who received at least one dose of study drug.
Arm/Group | Placebo IV | 350 mg Ramucirumab IV | Placebo SC | 350 mg Ramucirumab SC (1x2 mL) | 350 mg Ramucirumab SC (2x2 mL) | 350 mg Ramucirumab SC (2x1 mL) | 700 mg Ramucirumab SC (2x2 mL)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/12 | 0/7 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/7 | 1/12 | 0/7 | 1/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/3 | 4/7 | 1/12 | 3/7 | 2/7 | 5/7 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=3) | 350 mg Ramucirumab IV (N=7) | Placebo SC (N=12) | 350 mg Ramucirumab SC (1x2 mL) (N=7) | 350 mg Ramucirumab SC (2x2 mL) (N=7) | 350 mg Ramucirumab SC (2x1 mL) (N=7) | 700 mg Ramucirumab SC (2x2 mL) (N=7)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=3) | 350 mg Ramucirumab IV (N=7) | Placebo SC (N=12) | 350 mg Ramucirumab SC (1x2 mL) (N=7) | 350 mg Ramucirumab SC (2x2 mL) (N=7) | 350 mg Ramucirumab SC (2x1 mL) (N=7) | 700 mg Ramucirumab SC (2x2 mL) (N=7)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Lilly or Supplier shall publish, discuss, or release data emanating from a study without the other party's express written permission which shall not be unreasonably withheld. Nothing herein shall limit supplier's right to respond to legal inquiries.

DOCUMENTS (2):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT04495478/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT04495478/SAP_001.pdf